CLINICAL TRIAL: NCT03214874
Title: Randomized,Open Label,Balanced,Two Treatment, Four Period, Two Sequence, Single Oral Dose, Crossover, Replicate Study Under Fasting Conditions to Test Within Subject Variability of 20mg ER Torsemide and Demadex Tablets in Healthy Adults
Brief Title: Within Subject Variability Study of ER Torsemide 20 mg Tablet in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sarfez Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CLCD-058-15
Record Dates: First submitted 2017-07-08; First posted 2017-07-12 (Actual); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Congestive Heart Failure; Chronic Kidney Diseases
MeSH Terms: conditions — Heart Failure; Renal Insufficiency, Chronic | interventions — Torsemide; Tablets

STUDY DESIGN:
Intervention Model Description: Fully Replicate double-crossover
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Demadex 20mg Tablet (Active Comparator): Demadex (IR Torsemide) 20mg tablet once daily is the reference listed drug (RLD) and is marketed for decades to treat edema in Chronic Congestive Heart Failure (CHF) and Chronic Kidney Disease (CKD) patients
  Interventions: Drug: Demadex 20mg Tablet
- ER Torsemide 20mg Tablet (Experimental): ER Torsemide 20mg tablet once daily is is the new formulation that will release the active ingredient over an extended period
  Interventions: Drug: ER Torsemide 20mg Tablet

INTERVENTIONS:
Drug: Demadex 20mg Tablet — Immediate Release (IR) Torsemide
  Other Names: Torsemide
  Arms: Demadex 20mg Tablet
Drug: ER Torsemide 20mg Tablet — Extended Release Torsemide 20 mg tablet given once daily
  Other Names: ER Torsemide
  Arms: ER Torsemide 20mg Tablet

SUMMARY:
The study will evaluate the within-subject variability of 20mg ER torsemide as compared to 20mg IR torsemide (Demadex) in fully replicate double-crossover trial in healthy volunteers, who are consuming a high-salt diet (300 mmol/day). The study will also evaluate the effects of ER torsemide and IR torsemide on 24h sodium excretion and total urinary excretion.

DETAILED DESCRIPTION:
Immediate Release (IR) Torsemide is a highly effective natriuretic drug but its short duration of action is a major drawback, which allows significant post-dose sodium retention, and as consequence, limits salt loss in patients with heart failure, unless dietary salt intake is severely restricted. Extended Release (ER) torsemide is being developed to address the drawback by prolonging the duration of action to increase sodium excretion even in patients who consume high salt diet (300 mmol/day).

In addition, IR torsemide induces large and abrupt urination that, in some patients, causes incontinence, and as a result, compliance becomes challenging. ER torsemide is formulated to cause robust but gradual urination over an extended period to reduce accidental wetting and improve compliance.

In this study, ER torsemide is tested for within-subject variability in fully replicate design double-crossover trial in healthy volunteers who are on a 300 mmol/day sodium diet (high salt diet). The primary endpoint of the study is full pharmacokinetics measurements after a single dose of either ER torsemide or IR torsemide (Demadex). The secondary endpoints are 24h sodium excretion and total urinary excretion.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female, non-smoker, weight 50 kg for male and 45 kg for female, clinically acceptable laboratory profiles with ECG and chest X-ray performed within 6 months

Exclusion Criteria:

* participation in bioavailability/bioequivalence studies,
* history of drug abuse or alcohol dependence,
* history of allergies including drug allergies,
* known hypersensitivity to Torsemide or related drugs,
* presence of clinically significant disorder,
* systolic blood pressure <90 mm Hg or > 140 mm Hg diastolic blood pressure,
* history of incontinence,
* positive urine drug screening etc.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2017-06-19 (Actual); Primary Completion 2017-07-20 (Actual); Study Completion 2017-07-20 (Actual)

PRIMARY OUTCOMES:
Peak plasma concentration | 24 hour
  Peak tosremide plasma concentration (Cmax) (ng/ml)
Total plasma concentration | 24 hour
  Area under the plasma concentration versus time curve (AUC) (hr/ng/ml)
Urinary excretion | 24 hour
  Torsemide excretion in urine (microgram/min) over 24h post dose

SECONDARY OUTCOMES:
Urinary sodium excretion | 24 hour
  24h sodium (mmol/min)
Urine output | 24 hour
  24h total urinary output (l/day)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Wilcox, MD, PhD, Principal Investigator — Georgetown University
Locations (1):
- I.E.C. Consultants, Bangalore, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Murray MD, Deer MM, Ferguson JA, Dexter PR, Bennett SJ, Perkins SM, Smith FE, Lane KA, Adams LD, Tierney WM, Brater DC. Open-label randomized trial of torsemide compared with furosemide therapy for patients with heart failure. Am J Med. 2001 Nov;111(7):513-20. doi: 10.1016/s0002-9343(01)00903-2. PMID 11705426